CLINICAL TRIAL: NCT00044239
Title: The Characterization of Childhood Onset Obsessive Compulsive Disorder and the PANDAS Subgroup
Brief Title: Characterization of Childhood-Onset Obsessive-Compulsive Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020281; 02-M-0281
Record Dates: First submitted 2002-08-22; First posted 2002-08-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-18

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Tic Disorders; Neurophyschological; Immunology; Magnetic Resonance Imaging; Basal Ganglia; Obsessive-Compulsive Disorder; Children; Adolescents; Magnetic Resonance Spectroscopy; PANDAS (Pediatric Autoimmune Neuropsychiatric Disorders Associated d; Obsessive Compulsive Disorder; OCD; Healthy Volunteers; HV
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Tic Disorders; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections

SUMMARY:
The purpose of this study is to learn more about Obsessive-compulsive Disorder (OCD) in children. OCD usually has a slow onset, and symptoms that may remain at a stable level over time. A subset of children with OCD has a sudden onset and symptoms that fluctuate in severity over time. This study will also compare healthy children to those with OCD. This is an observational study; children who participate will not receive any new or experimental therapies.

OCD affects nearly 1% of the pediatric population. The symptoms of this illness can interrupt development, causing significant psychological distress and producing life-long impairments in social, academic, and occupational functioning. A subgroup of pediatric OCD has been designated by the acronym PANDAS (Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal Infections). This type of OCD is characterized by sudden symptom onset and a relapsing-remitting course of illness; exacerbation of symptoms occurs with scarlet fever or strep. throat infections. This study will identify factors that distinguish children with PANDAS OCD from children with non-PANDAS OCD, and will compare both groups to healthy children.

Children with OCD and their parents are screened with interviews and a review of the child's medical records. Participants have an initial evaluation that includes a psychiatric, physical and neuromotor exam, neuropsychological testing, psychological interviews, and a blood test. Structural magnetic resonance imaging (MRS) scans of the brain are also obtained. The MRS scan does not use radiation.

After the initial evaluation, children with OCD have follow-up visits every 6 weeks for 12 to 24 months. They are seen yearly for 8 years after the study. If they have a significant improvement or worsening of their symptoms, they are asked to make a maximum of two extra visits. Parents of OCD patients are called four times a year to discuss any changes in the child's condition between yearly visits. All participants have a 1-year follow-up visit upon study completion.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) affects nearly 1% of the pediatric population. The intrusive symptoms of this illness can interrupt normative development, causing significant psychological distress and producing life-long impairments in social, academic, and occupational functioning. Current research supports a neurobiologic model for OCD. Converging lines of evidence suggest that a post-infectious autoimmune-mediated process may be associated with the pathogenesis of some pediatric cases. This subgroup has been designated by the acronym, PANDAS (Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections). The abrupt symptom onset and relapsing-remitting course of illness characteristic of the PANDAS subgroup appears to define a distinct cohort of patients, in whom symptom exacerbations occur synchronously with Group A beta-hemolytic streptococcal (GABHS) infections.

We propose to perform prospective, longitudinal evaluations of a group of 72 children with recent onset OCD and 72 age-/sex-matched healthy volunteers. All children will undergo a comprehensive baseline assessment, including physical, neurological and psychiatric evaluations, neuropsychological testing, structural MRI and MRS scans, and laboratory assays. The children with OCD will be evaluated in the NIMH outpatient clinic at six-week intervals for a 28-month period to obtain prospective ratings of neuropsychiatric symptom severity, physical and neurological assessments, and anti-streptococcal antibody titers. At the end of the observation period, each OCD patient will be placed into a cohort based on the course of his or her symptoms: those displaying an acute onset and episodic course of OCD will be assigned to the "episodic" group, while those children with a gradual onset and stable course will comprise the "persistent" group. We hypothesize that the episodic group will have GABHS infections concurrent with their neuropsychiatric symptoms exacerbations and will meet criteria for the PANDAS subgroup. In contrast, children in the persistent group are not expected to have distinct periods of relapse nor a temporal association between GABHS infections and worsening of their symptoms. We expect that children in the PANDAS subgroup will demonstrate cross-reactive antibodies (antistreptococcal/antineuronal) during symptom exacerbations. At the conclusion of the study, we will perform group comparisons between the episodic OCD and persistent OCD cohorts, as well as between the patients and controls. The purpose of these comparisons is to identify baseline markers of membership in the PANDAS subgroup. The possibilities include distinctive HLA subtypes, quantitative differences in cytokines distribution, unique MRS chemical profiles, or a specific pattern of deficits on neuropsychological tests of basal ganglia function.

ELIGIBILITY:
* INCLUSION CRITERIA:

OCD Participants (N = 72)

1. Aged 4-12 years and living within a four-hour commute from NIH
2. Currently meet DSM-IV criteria for OCD.
3. Recent onset of symptoms (less than 6 months.)

Healthy Controls (N = 60-72)

1. Age and sex matched to ODC participants.
2. Must be free of current or past psychopathology.

EXCLUSION CRITERIA:

OCD Participants:

1. Diagnosis of schizophrenia, schizoaffective, bipolar, delusional, or psychotic disorder; autistic spectrum disorder or pervasive developmental disorder; neurologic disorder other than tics; or rheumatic fever.
2. Significant or unstable medical illness.
3. Full scale IQ less than 80.

Healthy Controls:

1. Full scale IQ less than 80.
2. Significant or unstable medical illness.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2002-08-20; Study Completion 2010-05-18

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arkansas, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida
  - Cornell University, New York, New York
  - Utah State University, Logan, Utah

REFERENCES:
- [Background] Rosenberg DR, Keshavan MS, O'Hearn KM, Dick EL, Bagwell WW, Seymour AB, Montrose DM, Pierri JN, Birmaher B. Frontostriatal measurement in treatment-naive children with obsessive-compulsive disorder. Arch Gen Psychiatry. 1997 Sep;54(9):824-30. doi: 10.1001/archpsyc.1997.01830210068007. PMID 9294373
- [Background] Snider LA, Lougee L, Slattery M, Grant P, Swedo SE. Antibiotic prophylaxis with azithromycin or penicillin for childhood-onset neuropsychiatric disorders. Biol Psychiatry. 2005 Apr 1;57(7):788-92. doi: 10.1016/j.biopsych.2004.12.035. PMID 15820236
- [Background] Saxena S, Brody AL, Schwartz JM, Baxter LR. Neuroimaging and frontal-subcortical circuitry in obsessive-compulsive disorder. Br J Psychiatry Suppl. 1998;(35):26-37. PMID 9829024